CLINICAL TRIAL: NCT05899686
Title: Effect of Tetanic Stimuli on Photoplethysmogram During General Anesthesia
Brief Title: Effect of Location of Tetanic Stimuli on Photoplethysmogram Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PT1502
Record Dates: First submitted 2023-05-06; First posted 2023-06-12 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stress Reaction
Keywords: photoplethysmography; stress response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Each participant will receive three tetanic stimuli. They are applied to the same three anatomical locations in each subject, but the order at which they are delivered to these locations will be random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tetanic Stimulus (Experimental): all participants receive the same intervention, which is three tetanic stimuli applied to three different anatomical locations. The three anatomical locations are identical in all subjects.
  Interventions: Device: Tetanic Stimulus

INTERVENTIONS:
Device: Tetanic Stimulus — 5 second 100 Hz 70 mA tetanic stimulus will be applied to three different anatomical locations in each subject.

SUMMARY:
The effect of the location of tetanic stimulus on photoplethysmography signals will be studied in patients under general anesthesia.

DETAILED DESCRIPTION:
A 5 second 100 Hz 70 mA tetanic stimulus will be applied to three different locations (Ulnar nerve, Facial nerve, Posterior Tibial nerve) in a random order in patients who are under general anesthesia. Tetanic stimuli are used routinely during general anesthesia to assess effectiveness of neuromuscular blockade. These tetanic stimuli are noxious stimuli that elicit a stress response which can be quantified using photoplethysmography. This study investigates if the magnitude of the tetanus induced stress response is dependent on the location of the tetanic stimulus as measured by photoplethysmography.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients
* Undergoing general anesthesia
* Able to consent in english
* 18 years of age or older

Exclusion Criteria:

* Under 18 years of age
* unable to consent in english
* receiving regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Talke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Principal investigator will provide data for reasonable requests

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stimuli were administered to three locations: A, B and C. Thus, there were 6 possible location sequences. ABC, ACB, BAC, BCA, CAB and CBA. These six location sequences were randomized in blocks of six (one of each) o that the sequence itself would not generate a bias. Thus, with 12 participants, each location sequence had two participants enrolled. For analysis the data for each location was pooled, independent of the location sequence.
Groups:
- Tetanic Stimulus: all participants receive the same intervention
  Tetanic Stimulus: 5 second 100 Hz 70 mA tetanic stimulus will be applied to each subject at three different anatomical locations. The order of the three locations will be randomized.
Period: Overall Study
Arm/Group | Tetanic Stimulus
Started | 12
Completed | 11
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Tetanic Stimulus: all participants receive the same intervention
  Tetanic Stimulus: 5 second 100 Hz 70 mA tetanic stimulus will be applied to three different locations in a random order
Arm/Group | Tetanic Stimulus
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tetanic Stimulus Induced Change in Photoplethysmography Light Transmission (in Analog to Digital Units as Measured Using a Pulse Oximeter) From Pre Stimulus Baseline
Description: Tetanic stimulation will induce peripheral vasoconstriction. This will be measured using photoplethysmography. During peripheral vasoconstriction the light transmission through finger will increase. The primary outcome will be the maximum change in light transmission (as measured by photoplethysmography) within 60 seconds after a tetanic stimulus as compared to pre stimulus baseline values. These maximal light transmission changes will be compared between the three different tetanic stimulus sites
Time Frame: Maximum light transmission change from pre tetanic stimulus baseline within 60 seconds after the tetanic stimulus
Measure: Mean (Standard Deviation); unit: percentage change from baseline value
Arm/Group | Tetanic Stimulus
Number analyzed (Participants) | 10
percentage change from baseline value
  Location 1 | -50 (19)
  Location 2 | -52 (18)
  Location 3 | -44 (19)
Statistical Analysis 1: Comparison: Tetanic Stimulus; Maximum percent change from baseline (light transmittance) during 60 heart beats after the tetanic stimulus were compared between the three stimulus locations using ANOVA; Test type: Equivalence — Equivalence was defined as ANOVA p<0.05; p = 0.65, ANOVA

ADVERSE EVENTS:
Time Frame: Principal investigator interviewed all subjects regarding adverse events after patients recovered from anesthesia, the day of the study.
Description: Principal investigator interviewed all subjects regarding adverse events after the surgical procedure and anesthesia.
Arm/Group | Tetanic Stimulus
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No